CLINICAL TRIAL: NCT02986256
Title: Comparative Study, Randomized in Parallel Groups, Evaluating the Consequences of the Management of Diabetic Foot Ulcers by Telemedicine Versus Conventional Monitoring on the Number of Hospital Days in Diabetic Patients
Brief Title: Evaluation of the Management of Diabetic Foot Ulcers by Telemedicine on the Number of Hospital Days in Diabetic Patients
Acronym: TELEPIED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-A01136-45
Record Dates: First submitted 2016-11-24; First posted 2016-12-08 (Estimated); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus; Ulcer Foot
Keywords: telemedicine
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventionnal Group (No Intervention): No intervention for this group. Patients will be followed by a usual care.
- "Telepied" Group (Experimental): Patients will be followed by a nurse referring to ulcers of the diabetic foot.
  Interventions: Behavioral: Taking pictures; Behavioral: Visit at home

INTERVENTIONS:
Behavioral: Taking pictures — Photograph of foot ulcer with transmission to referring nurse 1 time per week
  Arms: "Telepied" Group
Behavioral: Visit at home — Home visit by the referring nurse every 15 days
  Arms: "Telepied" Group

SUMMARY:
The TELEPIED project aims to show that it is possible to reduce the number of hospitalization days of a patient with ulcers of the foot thanks to a new organization of care, based on the intervention of a coordinating nurse interacting with the nurse in charge of the patient thanks to a telemedicine tool allowing the transfer of photos and ensuring itself a regular follow-up of the evolution of the wound and adapting the support nurse to the home if necessary.

It is a monocenter, randomized, in parallel study, in 180 diabetic patients with ulcers of the foot.

Patients included in the conventional group will be followed according to the usual practice Patients included in the "telepied" group will benefit from a personalized accompaniment by a nurse referring to diabetic foot ulcers who will guide and advise the nurse at home by acting by delegating tasks of the investigator.

The patient will be visited by the referring nurse every 15 days. During these visits, the referring nurse will have the objective to evaluate the evolution of the ulcer as well as the care performed. This visit also allows a close personalized accompaniment for the patient, who will benefit from an education adapted to the characteristics of ulcer (discharge modalities for example ..) and its way of life.

Every patients will be followed for one year (12 months).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Diabetic patients with foot ulcer
* Patient who agreed to participate in the study and sign free and informed consent
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Pregnant Woman
* Patient deprived of liberty by a judicial or administrative decision or a person subject to a legal protection measure
* Patient already involved in another clinical trial protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
Number of hospitalization days related to diabetic foot ulcers after one year of follow-up | 12 months

SECONDARY OUTCOMES:
Total direct care costs between the Telepied group and the control group | 12 months
  hospitalization costs, transport costs, nursing costs, liberal nursing costs, material costs, number of consultations with the doctor
Average duration of hospitalizations for an ulcer of the foot in the Telepied group versus the control group | 12 months
Ulcer recidivism rate in the Telepied group versus control group. | 12 months
Frequency of ulceration | 12 months
Duration of ulceration | 12 months
Healing rate between the Telepied group and the control group | 12 months
Amputation rate between the two groups | 12 months
Patient satisfaction score | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dured Dardari, MD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- Centre Hospitalier Sud-Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No